CLINICAL TRIAL: NCT00307775
Title: A Pilot Study to Examine the Efficacy of Vaginally Administered Oestradiol in the Treatment of Faecal Incontinence in Post Menopausal Women
Brief Title: Vaginal Estrogen for the Treatment of Faecal Incontinence in Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: London North West Healthcare NHS Trust (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06/VO1/6
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2007-02

CONDITIONS: Fecal Incontinence
Keywords: oestradiol, faecal incontinence, post menopausal; post menopausal women with faecal incontinence
MeSH Terms: conditions — Fecal Incontinence; Encopresis | interventions — Estradiol

INTERVENTIONS:
Drug: oestradiol

SUMMARY:
This study will address the following questions:

* Does the use of oestrogen inserted vaginally with an applicator, help with the symptoms of faecal (bowel) incontinence in women who are past the age of menopause?
* Do women find it easy to use?
* Is the treatment safe for the womb lining?
* Is there any systemic absorption of the treatment?

DETAILED DESCRIPTION:
Faecal incontinence affects about 5% of women, the most common cause is often cited by women as obstetric trauma. However in clinical practice many women report that their symptoms of faecal incontinence begin around the same time as menopause. A community survey examining the prevalence of faecal incontinence in menopausal women is in progress. If a correlation is found between the onset of menopause and the development of faecal incontinence, further investigation of effective treatment will be indicated.

The investigators want to investigate whether vaginally administered oestradiol can alleviate or improve symptoms in women who have faecal incontinence after the menopause. This is a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal women with faecal incontinence

Exclusion Criteria:

* No hormone replacement therapy (HRT) for at least 8 weeks prior to screening
* Diabetes mellitus
* Neurological disorder
* Terminal illness
* Current treatment for breast cancer
* Unable to give informed consent

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43
Dates: Start 2006-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Improvement of symptoms and quality of life (QoL) as measured by QoL questionnaires and physiological assessment

SECONDARY OUTCOMES:
Acceptance of treatment mode delivery, through questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Abernethy, RN ENB, Principal Investigator — London North West Healthcare NHS Trust; Joan Pitkin, MB BS BSc FRCS FRCOG, Study Chair — London North West Healthcare NHS Trust
Locations (1):
- North West London Hospitals NHS Trust, London, United Kingdom